CLINICAL TRIAL: NCT06155175
Title: Early Postoperative Non-steroidal Anti-inflammatory Drugs and Anastomotic Leakage for Rectal Cancer
Brief Title: Risk of NSAIDs on Anastomotic Leak for Rectal Surgery
Status: Completed | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Director, Third Military Medical University
Other Study IDs: 20230804
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Anastomotic Leak; Anti-Inflammatory Agents, Non-Steroidal
MeSH Terms: conditions — Anastomotic Leak | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSAIDs: patients were treated with NSAIDs postoperatively
  Interventions: Drug: NSAIDs
- No-NSAIDs: patients were not treated with NSAIDs postoperatively

INTERVENTIONS:
Drug: NSAIDs — The exposure to NSAIDs: NSAIDs was used at least once within the first day after surgery
  Groups: NSAIDs

SUMMARY:
Conflicting reports of the association between early postoperative non-steroidal anti-inflammatory drugs (NSAIDs) administration and anastomotic leak (AL) after rectal surgery have continued. The definition of AL and the exposure of NSAIDs differ from each other among studies, which may result in the different conclusions.

The aim of this retrospective study was to clarify the effect of NSAIDs on anastomotic leak from new angels.

DETAILED DESCRIPTION:
Concerning about the side effects induced by opioids, nonsteroidal anti-inflammatory drugs (NSAIDs) have gained its popularity in ERAS protocols. NSAIDs competitively inhibits the activity of cyclooxygenases (COXs), which are involved in migration of epithelial cell and mucosal restitution, angiogenesis and collagen synthesis during healing. Conflicting reports of the association between early postoperative non-steroidal anti-inflammatory drugs (NSAIDs) administration and anastomotic leak (AL) after rectal surgery have continued.

Notably, the definition of AL and the exposure of NSAIDs (i.e. NSAIDs administration) differ from each other among the studies, which may result in the different conclusions. In concrete terms, the definition of NSAIDs administration timing varies from the first day to the first week after surgery, while the AL was also defined in multiple ways (timing varies from 14 to 90 days postoperatively, or only leaks with operative intervention included). Most previous studies suggested that early and late AL are different entities with different risk factors. These interesting evidences indicate reconsidering the effect of NSAIDs on AL is needed.

Hence, investigators defined the NSAIDs administration as at least once in the early postoperative period--the day of and the day after surgery (NSAID group), to avoid the inclusion of patients started on NSAIDs secondary to a complication. At the same time, investigators also classified AL into early AL (confirmed within 6 days) and late AL (over 6 days). Moreover, concerning the higher rate of AL in rectal surgery than colonic surgery and the trend of minimally invasive surgery, investigators performed the current study, aiming to clarify the association between early postoperative NSAIDs and anastomotic leak in rectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven adenocarcinoma of the rectum
* Age over 18 years old
* Patients underwent non-emergency minimally invasive surgery with a primary anastomosis

Exclusion Criteria:

* Incomplete medical records
* Patients with distant metastasis before surgery
* Patients with multiple primary colorectal carcinomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent elective rectal resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 1969 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative anastomotic leak | within 30 days
  The primary outcome was anastomotic leak within 30 days after surgery. AL was defined as observing clinical signs of leak (such as high fever, abdominal pain, increasing of inflammatory factors in blood, purulent or fecal drainage from the drain, wound or vagina), and was confirmed by digital imaging or reoperation. Early AL was defined as being confirmed within 6 days postoperatively while late AL was defined as being confirmed after 6 days postoperatively

SECONDARY OUTCOMES:
The incidence of postoperative compolications | within 30 days
  Secondary outcomes include wound infection, anastomotic bleeding and obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: WeiDong Tong, MD, Study Director — Department of General Surgery, Daping Hospital, Army Medical University, Chongqing 400042, China
Locations (1):
- Army Medical Center, Chongqing, None Selected, China